CLINICAL TRIAL: NCT04380675
Title: Music Listening to Decrease Pain and Discomfort During Extracorporeal Shock Wave Lithotripsy (ESWL)
Brief Title: Music During ESWL for Entire Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Andrea Bosio, Principal investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOUCSSTURAB002
Record Dates: First submitted 2015-12-04; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Kidney Calculi; Lithotripsy; Pain Management; Music
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music during ESWL (Active Comparator): Patients listen to music during ESWL
  Interventions: Other: Music
- ESWL without music (No Intervention): Patients don't listen to music during ESWL

INTERVENTIONS:
Other: Music — Music listening during ESWL
  Arms: Music during ESWL

SUMMARY:
The aim of this study is to evaluate if music listening relieves pain and discomfort during Extracorporeal Shock-Waves Lithotripsy (ESWL).

DETAILED DESCRIPTION:
Patients undergoing ESWL and interested in music listening are randomly divided in two groups: patients in group A listen to music during the ESWL treatment, patients in group B do not.

At the end of the treatment patients are asked to fill in a questionnaire. They are asked if they were pleased to have had the opportunity to listen to music during ESWL, if they would like to listen to music again in case of further treatments, if they consider music helpful in relieving pain and discomfort during ESWL. Patients are also asked to mark their level of pain during each part of the treatment on a visual analogue scale (VAS) for pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ESWL and interested in music listening

Exclusion Criteria:

* Contraindication to ESWL
* No interest in music listening
* Age < 18 and > 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
change in VAS score | 10 mins after SWL treatment completed
  Visual analogue scale (VAS) - 0 to 10, higher values, worse pain

SECONDARY OUTCOMES:
change in Soundwave voltage (kV) | 10 mins after SWL treatment completed
  change in Soundwave voltage (kV)
change in analgesic request | 10 mins after SWL treatment completed
  change in analgesic request
change in requested interruptions | 10 mins after SWL treatment completed
  change in requested interruptions
change in Soundwave number | 10 mins after SWL treatment completed
  change in Soundwave number

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bosio, MD, Principal Investigator — AOU Città della Salute e della Scienza Torino
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Italy